CLINICAL TRIAL: NCT02490007
Title: Case-control Study of the Association Between Pertussis Vaccination in Infancy and the Risk of IgE-mediated Food Allergy
Brief Title: Pertussis Immunisation and Food Allergy
Acronym: PIFA
Status: Completed | Type: Observational
Sponsor: Telethon Kids Institute (Other)
Collaborators: Princess Margaret Hospital for Children (Other); Royal Children's Hospital (Other); Women's and Children's Hospital, Australia (Other Government); Sydney Children's Hospitals Network (Other); National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Other Study IDs: CVID/2015-02
Record Dates: First submitted 2015-06-30; First posted 2015-07-03 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2019-04

CONDITIONS: Food Allergy
Keywords: Acellular pertussis vaccine; whole cell pertussis vaccine; IgE-mediated food allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Allergy Cases: All participants appear on the Australian Childhood Immunisation Register (ACIR) and have received their first pertussis vaccination before the age of 16 weeks. They will have been born during the period of change over from whole cell pertussis vaccine to acellular pertussis vaccine (1997-1999). Allergy case participants have all attended allergy clinics associated with tertiary teaching hospitals. They have confirmed IgE-mediated food allergy as defined by the case description and as ascertained by their medical records.
- Controls: All participants appear on the Australian Childhood Immunisation Register (ACIR) and have received their first pertussis vaccination before the age of 16 weeks. They will have been born during the period of change over from whole cell pertussis vaccine to acellular pertussis vaccine (1997-1999).

SUMMARY:
Aim To assess the possible food allergy-preventive benefit of using whole cell pertussis(wP) vaccination compared with acelluar pertussis vaccine(aP) for whooping cough vaccination in childhood.

Background Whooping cough, caused by the bacteria, Bordetella pertussis, represents a significant public health burden in Australia and around the world. Acellular pertussis vaccination (aP) replaced whole cell vaccination against pertussis (wP) in the late 1990s. This replacement coincides temporally in an observed rapid rise in the occurrence of severe food allergy responses. Previous research has suggested that acellular pertussis vaccination results in the development of immunity that may predispose children to allergic responses. A retrospective case-controlled trial design, targeting cases of previously diagnosed allergy, and comparing case vaccination history to that of the whole population, is a powerful means of assessing the association between immunisation and allergy.

Participant Groups 1000 allergy cases, 10,000 controls

Project Design This is a retrospective individually-matched case-control study of Australian children born during the period of transition from use of wP vaccines to aP vaccines (year of birth 1997-1999 inclusive) and who are registered on the Australian Children Immunisation Register. Cases will be drawn from allergy clinics associated with tertiary teaching hospitals around Australia.

Methods Cases: will be retrospectively identified from patient lists from allergy clinics around Australia, born during the period of pertussis vaccine changeover, and be confirmed to have IgE-mediated food allergy on the basis of 1) a documented history of consistent clinical symptoms following ingestion of an implicated food, and 2) evidence of sensitisation to that food via laboratory testing.

Controls: Controls will be sampled from a de-identified database of children born during the transition from wP to aP vaccination appearing on the ACIR. Cases and controls will be matched by date of birth (+/-7 days), jurisdiction and socioeconomic decile.

Expected outcomes: Following the study, investigators will be able determine if there is an association between the type of vaccination received and development of IgE mediated food allergy. If whole cell vaccination is found to have a protective association against the development of allergy, this will have profound impact on health policy in Australia and around the world.

DETAILED DESCRIPTION:
BACKGROUND Atopic diseases have become the most important cause of chronic morbidity among children in wealthy countries. In particular, food allergy, including life-threatening food-related anaphylaxis, is growing at an alarming rate. For example, one Australian allergy clinic observed a 12-fold rise in consultations for food allergy in children between 1995 and 2006. In the 15 years to 2009/10, hospitalisations for food-related anaphylaxis in young Australian children increased more than 8-fold. No effective broadly implementable strategies to curb this 'second wave' of atopic disease have been discovered.

In Australia, an abrupt rise in food allergy coincided closely with the replacement of the antigenically complex whole-cell pertussis vaccine (wP) with the subunit acellular pertussis vaccine (aP) beginning in the late 1990s. Pertussis vaccine protects against Bordatella Pertussis, the causative agent of whooping cough.

Investigators previously shown the marked differences in the immune stimulating profile of wP compared with aP. wP has been shown to induce strong Th1 type immunity while aP induces a Th2 type response. Immune responses can be broadly grouped into cellular (Th1) and antibody mediated immunity (Th2). Natural protective immunity to pertussis relies on strong Th1 type responses to clear the pathogen. This is closely mimicked by the immunity induced by whole cell vaccine (wP). In contrast, the acellular vaccine relies on the development of antibody mediated protection. While antibody mediated responses are protective in the short term, the strong induction of Th2 responses may be deleterious to other aspects of the immune response.

The developing infant immune system has been shown to have a Th2 bias, which may be further skewed by the delivery of a vaccine with a strong Th2 immune profile. Dysregulation of the Th1/Th2 balance which should exist in the immune system can lead to disease states. Predominance of a Th2 environment leads to the development of atopy and allergy. A number of studies, exemplified by those from our centre, detail the Th2 immune bias induced in some infants who received DTaP-only schedules, resulting in excessive IgE production against vaccine antigens. This is likely due to the combined effect of 1) carry-over of the Th2-biased in utero phenotype, 2) the presence of alum and pertussis toxin which have Th2-adjuvantising properties, and 3) the absence of the balancing Th1-stimulating ligands present in DTwP. These effects manifest most strongly in infancy and among children with evidence of an underlying Th2-skewed phenotype.

Studies have demonstrated that the inclusion of even a single wP dose in a pertussis priming schedule is associated with a reduction in Th2-polarised T cell memory and the magnitude of the IgE response compared with a aP-only schedule. Based on these findings it is hypothesised that the inclusion of a single wP dose in the pertussis priming schedule might preserve the Th1/Th2 balance of the developing infant immune system.

Thus, this study will test the hypothesise that removal of wP from the infant vaccine schedule has contributed to the observed rise in IgE-mediated food allergy.

AIM To assess the possible food allergy-preventive benefit of using wP compared with aP for pertussis vaccination in childhood.

OBJECTIVES AND OUTCOME MEASURES

Primary objective To determine if Australian children born between 1997 to 1999 (inclusive) who received wP as their first pertussis vaccine dose in infancy were less likely to subsequently develop IgE-mediated food allergy compared with contemporaneous children who received aP as their first pertussis vaccine dose in infancy.

Secondary objectives To determine if Australian children born in the years 1997 to 1999 (inclusive) who received at least one dose of a wP pertussis vaccine at any age were less likely to subsequently develop IgE-mediated food allergy compared with contemporaneous children who received only aP pertussis vaccines.

To determine if Australian children born in the years 1997 to 1999 (inclusive) who received wP pertussis vaccines exclusively were less likely to subsequently develop IgE-mediated food allergy compared with contemporaneous children who received only aP pertussis vaccines.

STUDY DESIGN This is a retrospective individually-matched case-control study of Australian children born during the period of transition from use of wP containing pertussis vaccines to aP containing pertussis vaccines (year of birth 1997-1999 inclusive) and who are registered on ACIR and received their first dose of pertussis vaccine before age 16 weeks. Cases will be drawn from allergy clinics associated with tertiary teaching hospitals around Australia. 1000 cases, identified as having IgE mediated food allergy from reviewing case histories, and appearing on ACIR will be enrolled. Controls will be drawn from a de-identified database of the Australian Childhood Immunisation Register held by the National Centre for Immunisation Research and Surveillance of Vaccine Preventable Diseases. Each case will be individually matched to 10 controls.

Project coordination and epidemiological analysis will be conducted from the Wesfarmers Centre of Vaccines and Infectious Diseases at the Telethon Kids Institute Western Australia.

STATISTICS AND ANALYSIS Sample size and power considerations Sample size: A study with 1000 matched sets of cases and controls, with 10 matched controls for each case, will have at least 80% power to detect a 17% lower risk (odds ratio 0.83) of food allergy among children who received wP as their first dose of pertussis vaccine compared with those who received aP as their first dose. This assumes that: (i) 50% of controls receive a first pertussis vaccine dose of wP; (ii) the correlation coefficient for exposure (first dose of wP) between matched cases and controls is 0.5; and (iii) a significance level of 5% (α=0.05). Investigators believe that a small effect size will not influence policy or research direction. If only 500 cases meet the case criteria the study will still have at least 80% power to detect a 23% lower risk (odds ratio 0.77) of food allergy.

Description of Statistical Methods The cohort characteristics will be summarised by case or control status using means and standard deviations for symmetric distributions and medians and inter-quartile ranges for asymmetric distributions. Conditional logistic regression will be used to estimate odds ratios and the corresponding 95% confidence intervals for the associations between (exposure) pertussis vaccine type (wP or aP) and the risk of IgE-mediated food allergy. Because controls will be sampled from the register cohort irrespective of past or future case status, the odds ratio will be interpreted as an unbiased estimator of the relative risk of food allergy among children receiving wP compared with aP vaccines.

ELIGIBILITY:
Eligibility Criteria

1. All cases and controls must be registered on ACIR as having had a first dose of any pertussis containing vaccine before age 16 weeks and during the period of time in which the transition between aP and wP vaccine occurred; birth dates within 1st Janurary 1997 and 31st December 1999 depending on the jurisdiction.

Case Inclusion Criteria- Cases will be considered to have IgE-mediated food allergy on the basis of

1. a documented history of consistent clinical symptoms following ingestion of an implicated food, and
2. evidence of sensitisation to that food via either positive skin-prick test or elevated specific IgE to the implicated food, with onset after the first pertussis-containing vaccine but before age 15 years.

IgE-mediated food allergy is defined as BOTH:

1. The clinical notes or clinical letter arising from the allergy consult must explicitly document the presence of one or more of the following features. Onset of at least one these features must be within 1 hour of ingestion of suspected food where this can reasonably inferred from statements such as "immediate", "within x mins" where x is <60:

   * urticaria
   * angioedema
   * emesis
   * vocal hoarseness
   * persistent cough
   * wheeze
   * stridor
   * collapse
   * hypotension

   AND
2. Documented evidence of allergic sensitisation to the implicated food through EITHER:

   * specific IgE positive (serum specific IgE >0.35KU/l) to suspected food ), OR
   * positive skin prick test (wheal diameter >3mm) against suspected food (SPT) Evidence of sensitisation must be at the time of consultation or the 6 months after the clinical encounter for the case to meet definition.

Exclusion Criteria- none

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All participants appear on the Australian Childhood Immunisation Register (ACIR) and have received their first pertussis vaccination before the age of 16 weeks. They will have been born during the period of change over from whole cell pertussis vaccine to acellular pertussis vaccine (1997-1999). Allergy case participants have all attended allergy clinics associated with tertiary teaching hospitals. They have confirmed IgE-mediated food allergy as defined by the case description and as ascertained by their medical records.
Sampling Method: Non-Probability Sample
Enrollment: 508 (Actual)
Dates: Start 2015-10; Primary Completion 2018-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Diagnosis of IgE-mediated food allergy | birth-15 years
  To determine if children born between 1997 to 1999 who received wP as their first pertussis vaccine dose in infancy were less likely to develop IgE-mediated food allergy compared with children who received aP as their first pertussis vaccine dose

SECONDARY OUTCOMES:
Diagnosis of IgE-mediated food allergy | birth-15 years
  To determine if children born between 1997 to 1999 who received at least one dose of a wP pertussis vaccine at any age were less likely to develop IgE-mediated food allergy compared with children who received only aP pertussis vaccines. ACIR documented receipt of at least 1 dose of wP at any age with other doses as either wP, aP, or none OR only aP containing vaccines for all pertussis immunisations.
Diagnosis of IgE-mediated food allergy | birth-15 years
  To determine if Australian children born in the years 1997 to 1999 (inclusive) who received wP exclusively were less likely to subsequently develop IgE-mediated food allergy compared with contemporaneous children who received only aP pertussis vaccines. ACIR documented receipt of only wP containing vaccine for all pertussis immunisations or only aP containing vaccines for all pertussis immunisations.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Snelling, BMBS PhD, Principal Investigator — Telethon Kids Institute
Locations (1):
- Princess Margaret Childrens Hospital, Subiaco, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mullins RJ. Paediatric food allergy trends in a community-based specialist allergy practice, 1995-2006. Med J Aust. 2007 Jun 18;186(12):618-21. doi: 10.5694/j.1326-5377.2007.tb01077.x. PMID 17576175
- [Background] Torvaldsen S, Hull BP, McIntyre PB. Using the Australian Childhood Immunisation Register to track the transition from whole-cell to acellular pertussis vaccines. Commun Dis Intell Q Rep. 2002;26(4):581-3. doi: 10.33321/cdi.2002.26.60. PMID 12549528
- [Background] Mills KH, Ryan M, Mcguirk P, Griffin F, Murphy G, Mahon B. The immunology of bordetella pertussis infection. Biologicals. 1999 Jun;27(2):77. doi: 10.1006/biol.1999.0183. No abstract available. PMID 10600187
- [Background] Barlow WE, Davis RL, Glasser JW, Rhodes PH, Thompson RS, Mullooly JP, Black SB, Shinefield HR, Ward JI, Marcy SM, DeStefano F, Chen RT, Immanuel V, Pearson JA, Vadheim CM, Rebolledo V, Christakis D, Benson PJ, Lewis N; Centers for Disease Control and Prevention Vaccine Safety Datalink Working Group. The risk of seizures after receipt of whole-cell pertussis or measles, mumps, and rubella vaccine. N Engl J Med. 2001 Aug 30;345(9):656-61. doi: 10.1056/NEJMoa003077. PMID 11547719
- [Background] Feunou PF, Bertout J, Locht C. T- and B-cell-mediated protection induced by novel, live attenuated pertussis vaccine in mice. Cross protection against parapertussis. PLoS One. 2010 Apr 15;5(4):e10178. doi: 10.1371/journal.pone.0010178. PMID 20419113
- [Background] Mills KH, Ryan M, Ryan E, Mahon BP. A murine model in which protection correlates with pertussis vaccine efficacy in children reveals complementary roles for humoral and cell-mediated immunity in protection against Bordetella pertussis. Infect Immun. 1998 Feb;66(2):594-602. doi: 10.1128/IAI.66.2.594-602.1998. PMID 9453614
- [Background] Dannemann A, van Ree R, Kulig M, Bergmann RL, Bauer P, Forster J, Guggenmoos-Holzmann I, Aalberse RC, Wahn U. Specific IgE and IgG4 immune responses to tetanus and diphtheria toxoid in atopic and nonatopic children during the first two years of life. Int Arch Allergy Immunol. 1996 Nov;111(3):262-7. doi: 10.1159/000237376. PMID 8917121
- [Background] Rowe J, Macaubas C, Monger T, Holt BJ, Harvey J, Poolman JT, Loh R, Sly PD, Holt PG. Heterogeneity in diphtheria-tetanus-acellular pertussis vaccine-specific cellular immunity during infancy: relationship to variations in the kinetics of postnatal maturation of systemic th1 function. J Infect Dis. 2001 Jul 1;184(1):80-8. doi: 10.1086/320996. Epub 2001 May 29. PMID 11398113
- [Background] Rowe J, Yerkovich ST, Richmond P, Suriyaarachchi D, Fisher E, Feddema L, Loh R, Sly PD, Holt PG. Th2-associated local reactions to the acellular diphtheria-tetanus-pertussis vaccine in 4- to 6-year-old children. Infect Immun. 2005 Dec;73(12):8130-5. doi: 10.1128/IAI.73.12.8130-8135.2005. PMID 16299307
- [Background] Gruber C, Lau S, Dannemann A, Sommerfeld C, Wahn U, Aalberse RC. Down-regulation of IgE and IgG4 antibodies to tetanus toxoid and diphtheria toxoid by covaccination with cellular Bordetella pertussis vaccine. J Immunol. 2001 Aug 15;167(4):2411-7. doi: 10.4049/jimmunol.167.4.2411. PMID 11490032
- [Derived] Estcourt MJ, Marsh JA, Campbell DE, Gold MS, Allen KJ, Richmond P, Waddington CS, Snelling TL. Protocol for Pertussis Immunisation and Food Allergy (PIFA): a case-control study of the association between pertussis vaccination in infancy and the risk of IgE-mediated food allergy among Australian children. BMJ Open. 2018 Jan 31;8(1):e020232. doi: 10.1136/bmjopen-2017-020232. PMID 29391374

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT02490007/Prot_SAP_000.pdf